CLINICAL TRIAL: NCT00058019
Title: A Phase II Study of Epothilone B Analog BMS-247550 (NSC 710428) in Patients With Relapsed Aggressive Non-Hodgkin's Lymphomas
Brief Title: Ixabepilone in Treating Patients With Relapsed or Refractory Aggressive Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00031; NCI-2009-00031 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-5913; UCCRC-NCI-5913; CDR0000285683; UCCRC-11965B; 11965B (Other: University of Chicago); 5913 (Other: CTEP); P30CA014599 (NIH); N01CM62202 (NIH); N01CM62201 (NIH); NCT01660269 (obsolete NCT alias)
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Results first posted 2014-02-27 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2011-10

CONDITIONS: Anaplastic Large Cell Lymphoma; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Follicular; Lymphoma, Mantle-Cell | interventions — ixabepilone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (chemotherapy) (Experimental): Patients receive ixabepilone IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression, unacceptable toxicity, or if the patient becomes a candidate for stem cell transplantation.
  Interventions: Drug: ixabepilone

INTERVENTIONS:
Drug: ixabepilone — Given IV
  Other Names: BMS-247550; epothilone B lactam; Ixempra

SUMMARY:
This phase II trial is studying how well ixabepilone works in treating patients with relapsed or refractory aggressive non-Hodgkin's lymphoma. Drugs used in chemotherapy, such as ixabepilone, work in different ways to stop cancer cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the objective overall response rate of patients with relapsed or refractory aggressive non-Hodgkin's lymphoma treated with BMS-247550 (ixabepilone).

II. Determine the safety and toxicity of this drug in these patients. III. Determine the duration of response, overall survival, and time to progression in patients treated with this drug.

OUTLINE: This is a multi-center study.

Patients receive ixabepilone intravenously (IV) over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression, unacceptable toxicity, or if the patient becomes a candidate for stem cell transplantation.

Patients are followed every 8 weeks until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed aggressive non-Hodgkin's lymphoma of 1 of the following cellular types:

  * Grade III follicular center
  * Diffuse large B-cell
  * Mantle cell
  * Primary mediastinal B-cell
  * Burkitt's
  * High-grade B-cell (Burkitt-like)
  * Anaplastic large cell of 1 of the following subtypes:

    * CD30-positive
    * T-cell
    * Null cell
    * Hodgkin's-like
* Relapsed or refractory disease after prior standard chemotherapy, meeting criteria for 1of the following cohorts:

  * Cohort 1 (relapsed but chemosensitive): Prior complete response (CR) or partial response (PR) lasting at least 4 weeks after the most recent prior therapy
  * Cohort 2 (refractory): Stable disease or less than a PR after the most recent prior therapy

    * No progressive disease after the most recent prior therapy
* Measurable disease

  * At least 1 bidimensionally measurable lesion at least 10 mm by conventional techniques or clinical exam
* Ineligible for or unwilling to undergo hematopoietic stem cell transplantation

  * Patients requiring debulking prior to transplant allowed
* No known CNS involvement by lymphoma

  * Prior CNS disease that has been successfully treated in patients with relapsed disease exclusively outside of the CNS may be allowed by the principal investigator
* Performance status - ECOG 0-2
* More than 3 months
* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,200/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 mg/dL
* AST/ALT no greater than 2.5 times upper limit of normal
* Creatinine no greater than 1.5 mg/dL
* Creatinine clearance at least 60 mL/min
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior allergic reaction or hypersensitivity to compounds containing Cremophor EL or agents of similar chemical or biological composition to BMS-247550
* No peripheral neuropathy grade 2 or greater
* No other currently active malignancy except nonmelanoma skin cancer or carcinoma in situ of the cervix (previously treated malignancy allowed if considered to be at less than 30% risk of relapse)
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No other concurrent uncontrolled illness
* No colony-stimulating factors (CSFs) within 24 hours of study chemotherapy
* No CSFs during first course of study therapy
* No concurrent filgrastim-SD/01
* No concurrent immunotherapy
* See Disease Characteristics
* At least 4 weeks since prior cytotoxic chemotherapy (6 weeks for nitrosoureas or mitomycin)
* No other concurrent chemotherapy
* No concurrent hormonal therapy
* At least 4 weeks since prior radiotherapy
* No concurrent therapeutic radiotherapy
* At least 4 weeks since prior surgery
* Recovered from prior therapy
* At least 7 days since prior cimetidine
* No concurrent cimetidine
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents
* No other concurrent anticancer medications
* No concurrent unconventional therapies, food, or vitamin supplements containing Hypericum perforatum

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2003-02; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonali Smith, Principal Investigator — University of Chicago
Locations (2):
- United States (2):
  - University of Chicago, Chicago, Illinois
  - M D Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One patient never received treatment and was excluded from analysis.
Groups:
- Cohort 1 (Chemosensitive): Ixabepilone was administered intravenously at a dose of 20 mg/m^2 over 1 hour weekly on days 1,8, and 15 of a 28-day cycle. Cohort 1(Chemosensitive) enrolled patients with a complete response or partial response lasting at least 4 weeks to their most recent therapy.
- Cohort 2 (Chmoresistant): Ixabepilone was administered intravenously at a dose of 20 mg/m^2 over 1 hour weekly on days 1,8, and 15 of a 28-day cycle. Cohort 2(Chemoresistant) enrolled patients with stable disease but less than a partial response to their most recent therapy.
Period: Overall Study
Arm/Group | Cohort 1 (Chemosensitive) | Cohort 2 (Chmoresistant)
Started | 39 | 12
Completed | 39 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Chemosensitive) | Cohort 2 (Chmoresistant) | Total
Number analyzed (Participants) | 39 | 12 | 51
Age, Continuous [Median (Full Range); unit: years] | 64 [44 to 90] | 73 [53 to 87] | 66 [44 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 5 | 17
  Male | 27 | 7 | 34
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 34 | 12 | 46
  African American | 1 | 0 | 1
  Hispanic | 4 | 0 | 4
LDH elevation [Number; unit: Participants]
  Yes | 16 | 6 | 22
  No | 23 | 6 | 29
Prior therapies [Number; unit: Participants]
  1 | 10 | 4 | 14
  2-3 | 17 | 5 | 22
  4 or more | 12 | 3 | 15
Prior rituximab [Number; unit: Participants]
  Yes | 34 | 11 | 45
  No | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Objective Overall Response Rate
Description: The 1999 international response criteria (http://www.ncbi.nlm.nih.gov/pubmed/10561185) as published by Cheson was used for the definition of target lesions and CT scans were used for response assessment. CR(complete response)/CRu(unconfirmed complete response) requires disappearance of all target lesions; PR (partial response) requires >=50% decrease in the sum of the products of the greatest diameters; Overall Response (OR)=CR/CRu+PR.
Time Frame: up to 3 years
Measure: Number; unit: participants
Arm/Group | Cohort 1 (Chemosensitive) | Cohort 2 (Chmoresistant)
Number analyzed (Participants) | 39 | 12
participants | 14 | 0
Statistical Analysis 1: Comparison: Cohort 1 (Chemosensitive) vs Cohort 2 (Chmoresistant); Test type: Superiority or Other; p = 0.022, Fisher Exact

2. Primary Outcome: Safety and Toxicity of Ixabepilone
Description: Number of patients experiencing adverse event grade 3 or above. Grade was determined by the National Cancer Institute Common Toxicity Criteria (CTC) version 2.0. Adverse events possibly, probably, or definitely attributed to use of ixabepilone.
Time Frame: up to 3 years
Measure: Number; unit: participants
Arm/Group | Cohort 1 (Chemosensitive) | Cohort 2 (Chmoresistant)
Number analyzed (Participants) | 39 | 12
participants | 27 | 8
Statistical Analysis 1: Comparison: Cohort 1 (Chemosensitive) vs Cohort 2 (Chmoresistant); Test type: Superiority or Other; p = 1.00, Fisher Exact

3. Secondary Outcome: Duration of Response
Description: Duration of response was measured from the time measurement criteria are met for CR(complete response)/CRu(unconfirmed complete response)/PR(partial response), whichever was first recorded, until the first date that PD(progressive disease) was objectively documented. According to the 1999 international response criteria as published by Cheson, CR/CRu is defined as the disappearance of all target lesions; PR is defined as >=50% decrease in the sum of the products of the greatest diameters; PD is defined as >=50% increase from nadir in the sum of the products of the greatest diameters of any previously identified abnormal node for PRs or nonresponders, or appearance of any new lesion during or at the end of therapy.
Time Frame: up to 3 years
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Cohort 1 (Chemosensitive) | Cohort 2 (Chmoresistant)
Number analyzed (Participants) | 14 | 0
Days | 291 [162 to NA] — The upper limit of 95% CI is undetermined because never drops below -1.96 due to the heavy censoring. |

4. Secondary Outcome: Overall Survival
Description: Defined as the time from the first day of therapy to the date of death. If the patient was lost to follow-up, survival was censored on the last date the patient was known to be alive.
Time Frame: up to 3 years
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Cohort 1 (Chemosensitive) | Cohort 2 (Chmoresistant)
Number analyzed (Participants) | 39 | 12
Days | 501 [340 to NA] — The upper limit of 95% CI is undetermined because never drops below -1.96 due to the heavy censoring. | 98 [67 to NA] — The upper limit of 95% CI is undetermined because never drops below -1.96 due to the heavy censoring.
Statistical Analysis 1: Comparison: Cohort 1 (Chemosensitive) vs Cohort 2 (Chmoresistant); Test type: Superiority or Other; p = 0.695, Log Rank

5. Secondary Outcome: Time to Progression
Description: Defined as the time from the first day of treatment until the date PD(progressive disease) or death is first reported. Patients who died without a reported prior progression was considered to have progressed on the day of their death. Patients who did not progress was censored at the day of their last tumor assessment. According to the 1999 international response criteria as published by Cheson, progression/progressive disease is defined as >=50% increase from nadir in the sum of the products of the greatest diameters of any previously identified abnormal node for PRs or nonresponders, or appearance of any new lesion during or at the end of therapy.
Time Frame: up to 3 years
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Cohort 1 (Chemosensitive) | Cohort 2 (Chmoresistant)
Number analyzed (Participants) | 39 | 12
Days | 112 [56 to 340] | 84 [67 to NA] — The upper limit of 95% CI is undetermined because never drops below -1.96 due to the heavy censoring.
Statistical Analysis 1: Comparison: Cohort 1 (Chemosensitive) vs Cohort 2 (Chmoresistant); Test type: Superiority or Other; p = 0.55, Log Rank

ADVERSE EVENTS:
Description: Adverse events possibly, probably, or definitely attributed to use of ixabepilone. The Adverse event report includes all patients experiencing adverse events with any grade while one of the primary outcomes (safety and toxicity of Ixabepilone) targeted patients experiencing adverse event grade 3 or above.
Arm/Group | Ixabeilone for Relapsed Aggressive NHL
Serious Adverse Events (participants affected / at risk) | 11/51
Other Adverse Events (participants affected / at risk) | 48/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabeilone for Relapsed Aggressive NHL (N=51)
Dehydration (Metabolism and nutrition disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 2
Lung infection (Infections and infestations) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neutrophil count decreased (Investigations) | 2
Palpitations (Cardiac disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Thromboembolic event (Vascular disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabeilone for Relapsed Aggressive NHL (N=51)
Peripheral sensory neuropathy (Nervous system disorders) | 32
Fatigue (General disorders) | 31
White blood cell decreased (Investigations) | 30
Nausea (Gastrointestinal disorders) | 24
Anemia (Blood and lymphatic system disorders) | 26
Hyperglycemia (Metabolism and nutrition disorders) | 8
Diarrhea (Gastrointestinal disorders) | 18
Platelet count decreased (Investigations) | 19
Neutrophil count decreased (Investigations) | 21
Anorexia (Metabolism and nutrition disorders) | 15
Constipation (Gastrointestinal disorders) | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 13
Lymphocyte count decreased (Investigations) | 13
Alopecia (Skin and subcutaneous tissue disorders) | 11
Aspartate aminotransferase increased (Investigations) | 9
Edema limbs (General disorders) | 3
Vomiting (Gastrointestinal disorders) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Alanine aminotransferase increased (Investigations) | 6
Hypocalcemia (Metabolism and nutrition disorders) | 4
Infections and infestations - Other, specify (Infections and infestations) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Dizziness (Nervous system disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
Weight loss (Investigations) | 4
Peripheral motor neuropathy (Nervous system disorders) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 3
Pain (General disorders) | 4
Alkaline phosphatase increased (Investigations) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 3
Fever (General disorders) | 4
Dysgeusia (Nervous system disorders) | 5
Injection site reaction (General disorders) | 4
Hyperkalemia (Metabolism and nutrition disorders) | 4
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Creatinine increased (Investigations) | 3
Dehydration (Metabolism and nutrition disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less